CLINICAL TRIAL: NCT07274657
Title: Superb Microvascular Imaging (SMI) and Two-Dimensional Endoscopic Ultrasound Guided Shear Wave Elastography (2D-SWE-EUS) in Differential Diagnosis of Pancreatic Adenocarcinoma (PA) From Other Pancreatic Solid Lesions (PSLs) and Pancreatic neuroendocrinE Tumors (pNETs) Malignancy
Acronym: SMILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-A01725-44
Record Dates: First submitted 2025-11-23; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Adenocarcinoma (MSI-H); Pancreatic Neuroendocrine Tumors (pNET)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New imaging arm (Experimental): New imaging arm involves characterization and diagnosis of PA and pNETs malignancy, using the linear-array EUS scope UCT-180 Olympus and the new Aplio i800 EUS Unit (Canon Olympus - CE marked) equipped with a SMI and 2D-SWE modes
  Interventions: Device: SMI and 2D-SWE modes

INTERVENTIONS:
Device: SMI and 2D-SWE modes — SMI and 2D-SWE are new imaging modes on the new Aplio i800 EUS Unit (Canon Olympus - CE marked)

SUMMARY:
Pancreatic adenocarcinoma (PA) is the most common tumor of the pancreas. Given its poor prognosis and the major therapeutic consequences, the discrimination between PA and other pancreatic solid lesions is mandatory.

Endoscopic ultrasound (EUS) is admitted as the most sensitive imaging procedure for the detection and characterization of pancreatic tumors. Over the past 30 years, EUS-guided tissue acquisition (EUS-TA), or more recently fine needle biopsy (EUS-FNB), has demonstrated its efficiency for tissue sampling and remains the gold standard for the pathologic diagnosis of pancreatic lesions.

The assessment of pancreatic tumor enhancement using ultrasound contrast agents (UCAs) in real time with imaging specific methods seems useful to improve their characterization either by contrast-enhanced EUS (CE-EUS) or, more recently, by contrast-harmonic EUS (CH-EUS). CH-EUS was already demonstrated useful to differentiate pancreatic adenocarcinoma from other pancreatic lesions.

EUS-Elastography (EUS-E) is another EUS image enhancement technique, which rational based on the difference in elasticity between the tissues. There are two types of elastographies: strain elastography (SE) and shear wave elastography (SWE). SE has proved useful for the characterization of pancreatic lesions and lymph nodes. However, this technique was demonstrated difficult to perform with adequate accuracy and reproducibility for pancreatic lesions and have many limitations. In some recent publications SWE was demonstrated moderate reliability.

Pancreatic neuroendocrine tumors (pNETs) are rare tumors, but according to the last epidemiological data, their incidence and prevalence are steadily rising.

Surgical resection is generally performed for pNETs due to their malignant potential. However, with increasing use of high-resolution conventional imaging, the significant incidence of small (≤ 2 cm) pancreatic neuroendocrine incidentaloma (pNET) has risen in recent decades.

EUS is recognized as the most sensitive procedure for the detection and characterization of pNETs. Overall sensitivity of EUS-TA for the diagnosis of pNETs is high, reaching 95.1% in recently published study, appearing higher in small lesions (≤ 20 mm) than in large lesions (> 20 mm).

The overall concordance rate for EUS-TA and surgical specimens grading varies from 58% to 86.4% and is higher for lesions ≤ 10 mm, 10-20 mm, comparing to lesions > 20 mm. These results confirm the risk of under or over-grading of pNETs on the EUS-TA specimen, independently of the needle size which used for the TA.

CH-EUS was also demonstrated accurate in the prediction of pNETs malignancy and useful for decision-making management of these tumors.

Hypothesis

Two new image enhancement EUS technologies were recently developed, able to assess precisely tumor microvascular density and the stiffness of pancreatic lesions, that is correlated to tumor's stroma fibrosis, and thus help to characterize and predict the malignancy, and accordingly, the management of the pancreatic solid lesions. It's particularly useful in overcoming EUS false-negative cases of PA and small pNETs malignancy diagnosis.

Superb Microvascular Imaging (SMI) is a novel doppler technique that enhances the range of visible blood flow, by revealing low velocity microvascular flow, enabling the capture of a higher-quality microvascular flow images. Based on the same principle as CH-EUS, which assesses tumor microvascularization, this technique is expected to be also useful for the PSLs malignancy diagnosis.

Shear Wave Elastography (SWE) relies on the properties of shear-wave propagation to offer an advanced assessment of their velocity

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PA) diagnosis

Pancreatic adenocarcinoma (PA) is the most common tumor of the pancreas, representing more than 90% of all solid pancreatic neoplasia and 55% -73% of solid pancreatic masses. Given its poor prognosis and the major therapeutic consequences, the discrimination between PA and other pancreatic solid lesions is mandatory.

Endoscopic ultrasound (EUS) is admitted as the most sensitive imaging procedure for the detection and characterization of pancreatic tumors. Based on only endosonographic features, it remains difficult to differentiate PA from other solid masses, the specificity (Spe) and accuracy of EUS for the diagnosis of pancreatic tumor malignancy range from 53-69% and 72-83%, respectively.

Over the past 30 years, EUS-guided tissue acquisition (EUS-TA), or more recently fine needle biopsy (EUS-FNB), has demonstrated its efficiency for tissue sampling and remains the gold standard for the pathologic diagnosis of pancreatic lesions.

Although several prospective randomized studies and meta-analyses have shown that FNB needles are significantly superior to FNA needles for the diagnosis of solid pancreatic tumors, the overall accuracy remains insufficient to rule out malignancy. Additional diagnostic criteria are then required.

The assessment of pancreatic tumor enhancement using ultrasound contrast agents (UCAs) in real time with imaging specific methods seems useful to improve their characterization either by contrast-enhanced EUS (CE-EUS) or, more recently, by contrast-harmonic EUS (CH-EUS). Contrast harmonic EUS (CH-EUS), was already demonstrated useful to differentiate pancreatic adenocarcinoma from other pancreatic lesions.

EUS-Elastography (EUS-E) is another EUS image enhancement technique, which rational based on the difference in elasticity between the tissues. There are two types of elastographies: strain elastography (SE) and shear wave elastography (SWE). Strain elastography has proved useful for the characterization of pancreatic lesions and lymph nodes. However, this technique was demonstrated difficult to perform with adequate accuracy and reproducibility for pancreatic lesions and have many limitations. In some recent publications SWE was demonstrated moderate reliability.

Pancreatic neuroendocrine tumors (pNETs)

Pancreatic neuroendocrine tumors (pNETs) are rare tumors, but according to the last epidemiological data, their incidence and prevalence are steadily rising.

Surgical resection is generally performed for pNETs due to their malignant potential. However, with increasing use of high-resolution conventional imaging, the significant incidence of small (≤ 2 cm) pancreatic neuroendocrine incidentaloma (pNET) has risen in recent decades. Given their unknown natural history due to the lack of literature, the significant morbidity and mortality of pancreatic surgery, the current French and European Neuroendocrine Tumor Society (ENETS) Guidelines suggests that conservative management may also be considered for the small size (≤ 2 cm) nonfunctional, asymptomatic and without criteria for malignancy pNETs, classified as G1 or low G2 according to the 2019 World Health Organization (WHO) classification system lesion, after multidisciplinary discussion and patient counseling.

EUS is recognized as the most sensitive procedure for the detection and characterization of pNETs. Overall sensitivity of EUS-TA for the diagnosis of pNETs is high, reaching 95.1% in recently published study, appearing higher in small lesions (≤ 20 mm) than in large lesions (> 20 mm).

The overall concordance rate for EUS-TA and surgical specimens grading varies from 58% to 86.4% and is higher for lesions ≤ 10 mm, 10-20 mm, comparing to lesions > 20 mm. These results confirm the risk of under or over-grading of pNETs on the EUS-TA specimen, independently of the needle size which used for the TA.

CH-EUS was also demonstrated accurate in the prediction of pNETs malignancy and useful for decision-making management of these tumors.

Hypothesis

Two new image enhancement EUS technologies were recently developed, able to assess precisely tumor microvascular density and the stiffness of pancreatic lesions, that is correlated to tumor's stroma fibrosis, and thus help to characterize and predict the malignancy, and accordingly, the management of the pancreatic solid lesions. It's particularly useful in overcoming EUS false-negative cases of PA and small pNETs malignancy diagnosis.

Superb Microvascular Imaging (SMI) is a novel doppler technique that enhances the range of visible blood flow, by revealing low velocity microvascular flow, enabling the capture of a higher-quality microvascular flow images. Based on the same principle as CH-EUS, which assesses tumor microvascularization, this technique is expected to be also useful for the PSLs malignancy diagnosis.

Shear Wave Elastography (SWE) relies on the properties of shear-wave propagation to offer an advanced assessment of their velocity and tissue elasticity, presenting the results quantitatively in a dynamic display.

The new developed image enhancement EUS technologies, SMI and 2D-SWE-EUS now available on the new Aplio i800 EUS unit (Canon-Olympus).

Given the lack of published data in the literature regarding the utility of SMI and 2D-SWE-EUS, it is essential to assess the performance of these two techniques in the differential diagnosis of SPLs and pNETs malignancy

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, age ≥ 18 years old
* Patient with diagnosed pancreatic solid or mixed (cystic component ≤25 % of tumor volume) lesion
* Patient with adequate understanding of written and spoken French, able to sign written informed consent
* Patient affiliated with a social security system

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient with usual contraindications to EUS- TA
* Patient with usual contraindications to SonoVue® administration
* Patient with a genetic syndrome associated pancreatic lesion (multiple neuroendocrine neoplasia type 1 (MEN1), type 1 neurofibromatosis (NF), Von-Hippel Lindau (VHL) disease)
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Patient unable to perform the monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Independent sensitivity assessment of each imaging technique, EUS-SMI, 2D-SWE-EUS and CH-EUS, according to final histopathological diagnosis for the diagnostic of PA | 12 months after EUS (Endoscopic ultrasound)-guided tissue acquisition (EUS-TA)
  Sensitivity is defined as the number of true positives (positive diagnoses in patients with PA) divided by the total number of patients with PA. The presence or absence of PA will be revealed by a final diagnosis based on:
  - The cyto-pathological result obtained by EUS-TA of the pancreatic lesion or the histo-pathological result obtained by surgery (if performed).
  And
  - Clinical follow-up data for 12 months: doubling in size of the primary tumor during the follow-up and/or vascular invasion and/or appearance of lymph nodes and/or distant metastases

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No